CLINICAL TRIAL: NCT03707613
Title: Learning Curve of Double-wire Cannulation Technique During Endoscopic Retrograde Cholangiopancreatography(ERCP): a Pilot Study
Brief Title: Learning Curve of Double-wire Cannulation Technique During Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associate Professor, Air Force Military Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KY20180081-3
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Biliary Cannulation; Endoscopic Retrograde Cholangiopancreatography
Keywords: ERCP; double guidewire technique; learning curve

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DWT learning curve (Experimental): Initial cannulation is performed with a wire-guided sphincterotome by a trainee. If the cannulation proves difficult (cannulation time >10min, cannulation attemtps >5 or inadvertent PD cannulation >1) and PD is inadvertently entered, DWT will be performed by one of the two trainees. If DWT fails within 5min or 5 attempts, a trainer will take over and continue the cannulation. To prevent PEP, all patients receive prophylactic PD stent and post-ERCP rectal indomethacin. Aggressive hydartion will be administrated at the discretion of endoscopists.
  Interventions: Procedure: DWT learning curve

INTERVENTIONS:
Procedure: DWT learning curve — trainees learn to perform DWT after unsuccessful initial cannulation

SUMMARY:
Selective cannulation is considered the most challenging step for most of endoscopic retrograde cholangiopancreatography (ERCP). Wire-guided cannulation is the standard technique for initial cannulation. When meeting difficulty, double wire technique (DWT) is widely used. With one guidewire occupying pancreatic duct(PD) , the following cannulation of CBD with a sphincterome preloaded with another guidewire often becomes feasible.

When performing DWT, a sphincterotome should enter the common duct of papilla through a small orifice and be placed in the left and upper direction of PD guidewire. Then another guidewire can be advanced into bile duct. As an advanced cannulation technique, DWT can be successfully performed in up to 80% of difficult patients. However, it can be technically difficult, especially for trainees or endoscopists without adequate experience.

Here we planned to prospectively record the procedures of double-wire cannulation by two trainees without prior experience of DWT. This study aims to delinate the learning curve of DWT and its safety by trainees.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-90 with native papilla
* patients with diffcult cannulation of bile duct
* Inadvertent pancreatic duct cannulation

Exclusion Criteria:

* Contraindications of ERCP
* Major or minor pancreatic duct as the targeted duct
* Prior EST or needle-knife precut before DWT
* Surgically altered gastrointestinal anatomy
* Papillary carcinoma or stone impaction within papilla
* Complete pancreas divisum
* Pregnant or breastfeeding women
* Unwilling or inability to provide consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Successful cannulation of bile duct within 5min or 5 attempts of cannulation | 3 hours
  It was defined by assurance of entering bile duct through cholangiogram during fluoroscopy.

SECONDARY OUTCOMES:
Successful cannulation time with DWT by trainees | 3 hours
  Successful cannulation time was defined by the time taken from the begining of DWT to entering bile duct successfully
Cannulation attempts with DWT by trainees | 3 hours
  One cannulation attempt was defined by touching papilla for more than 5 seconds.
Precut rate | 3 hours
  Precut includes the procedure of cannulation involving needle knife or dual knife and transpancreatic precut by a sphincterotome.
post-ERCP pancreatitis(PEP) | 48 hours
  PEP is defined according to Cotton's criteria. The severity classification is based on revised Atlanta criteria.
Overall ERCP-related complications | 48 hours
  Overall ERCP-related complations include PEP, bleeding, perforation, cholangitis and others, which is defined by Cotton's criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Ren G, Xi Y, Luo H, Liang S, Wang B, Tao Q, Luo B, Qin Q, Farrell JJ, Guo X, Wu K, Pan Y. Learning curve of double-guidewire technique by trainees during hands-on endoscopic retrograde cholangiopancreatography training. J Gastroenterol Hepatol. 2020 Dec;35(12):2176-2183. doi: 10.1111/jgh.15120. Epub 2020 Jun 23. PMID 32473040